CLINICAL TRIAL: NCT05030545
Title: Cardiovascular Manifestations of MR Activation in Primary Aldosteronism: Pilot Clinical Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jenifer M. Brown, M.D., Instructor in Medicine, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021P002400
Record Dates: First submitted 2021-08-26; First posted 2021-09-01 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Primary Aldosteronism; Hypertension
MeSH Terms: conditions — Hyperaldosteronism; Hypertension | interventions — Eplerenone; Mineralocorticoid Receptor Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Eplerenone Treatment (Experimental): Eplerenone (50-100mg daily, as tolerated by blood pressure and potassium) for 6 months
  Interventions: Drug: Eplerenone

INTERVENTIONS:
Drug: Eplerenone — After baseline cardiac imaging with PET and echocardiogram, participants will be treated with eplerenone for 6 months at a starting dose of 50mg daily and up to a maximally tolerated dose of 100mg daily, followed by repeat imaging with PET and echocardiogram.
  Other Names: Inspra; Mineralocorticoid Receptor Antagonist

SUMMARY:
This research study aims to learn more about the impact the hormone aldosterone on the heart. Primary aldosteronism is a condition where the body's adrenal glands make too much of the hormone aldosterone, which can cause high blood pressure and increase the risk of heart and kidney disease. Treatment with medications that block aldosterone can reduce that risk. This study is trying to learn whether treatment with a medication that blocks aldosterone can improve heart function in people who make too much aldosterone.

DETAILED DESCRIPTION:
The study evaluates the impact of 6 months of treatment with the mineralocorticoid receptor blocking medication eplerenone on the heart's blood flow, using a cardiac PET stress test, and on the heart's structure and function by echocardiogram.

Participants with a confirmed diagnosis of primary aldosteronism will undergo echocardiogram and cardiac PET stress test before and after 6 months of eplerenone treatment.

Participants without a confirmed diagnosis of primary aldosteronism but with hypertension and a recent clinical PET test and echocardiogram will undergo testing to make the diagnosis of primary aldosteronism. Those who test positive will go on to treatment with eplerenone for 6 months, followed by a cardiac PET scan and echocardiogram.

ELIGIBILITY:
Cohort A: Overt & Diagnosed PA

Inclusion Criteria:

* Adults aged 18-85
* Able to provide informed consent and willing to comply with the study
* Able to fit safely in PET/CT scanner (weight limit 500 pounds; diameter and circumference of PET/CT scanner are 70 cm and 220 cm, respectively)
* Hypertension treated with at least one antihypertensive drug
* Cohort A: Clinically confirmed diagnosis of PA not yet treated with mineralocorticoid receptor antagonists

Exclusion Criteria:

* History of MI, CABG, known cardiomyopathy (EF <40%, hypertrophic cardiomyopathy, and/or amyloid), cardiac transplantation
* Contraindication or allergy to eplerenone or spironolactone
* Current pregnancy or breastfeeding
* eGFR < 45 mL/min/1.73m2 or potassium > 5.1 on labs within the preceding 3 months
* Cohort A: Planned adrenalectomy in the subsequent 6 months

Cohort B: Subclinical & Undiagnosed PA

Inclusion Criteria:

* Adults aged 18-85
* Able to provide informed consent and willing to comply with the study
* Able to fit safely in PET/CT scanner (weight limit 500 pounds; diameter and circumference of PET/CT scanner are 70 cm and 220 cm, respectively)
* Hypertension treated with at least one antihypertensive drug
* Cohort B: Clinically indicated cardiac PET perfusion scan within the preceding 3 months and echocardiogram within the preceding 6 months

Exclusion Criteria:

* History of MI, CABG, known cardiomyopathy (EF <40%, hypertrophic cardiomyopathy, and/or amyloid), cardiac transplantation
* Contraindication or allergy to eplerenone or spironolactone
* Current pregnancy or breastfeeding
* eGFR < 45 mL/min/1.73m2 or potassium > 5.1 on labs within the preceding 3 months
* Cohort B: 10% or greater burden of ischemia on qualifying PET
* Cohort B: Planned coronary angiogram/revascularization in the subsequent 6 months.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in myocardial flow reserve (MFR, unitless ratio) | 6 months
  The primary outcome is to evaluate the change in MFR, as measured by PET, pre- vs post-6 months of eplerenone therapy

SECONDARY OUTCOMES:
Change in peak-stress myocardial blood flow (ml/min/g) | 6 months
  Peak stress myocardial blood flow is measured by PET after vasodilator-induced maximal hyperemia, before and after 6 months of eplerenone treatment
Change in Global Longitudinal Strain (%) | 6 months
  Global Longitudinal Strain is measured by echocardiography before and after 6 months of eplerenone treatment
Change in LV Mass Index (g/m2 of body surface area) | 6 months
  LV Mass Index is measured by echocardiography before and after 6 months of eplerenone treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No